CLINICAL TRIAL: NCT00832897
Title: "Evaluation of Topical Riboflavin Exposed to UVA Radiation and Implantation of Intrastromal Corneal Ring for Treatment of Keratoconus and Others Irregulars Astigmatisms."
Brief Title: Evaluation of Topical Riboflavin Exposed to UVA Radiation and Implantation of Corneal Ring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Federal University of São Paulo, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1915/07
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Keratoconus
Keywords: Keratoconus; riboflavin; cornea; crosslinking
MeSH Terms: conditions — Keratoconus; Corneal Diseases | interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eyedrop (Sham Comparator)
  Interventions: Procedure: Corneal collagen crosslinking
- Crosslinking (Active Comparator): The patients will be submitted to corneal collagen crosslinking, by use riboflavin eyedrop with UVA light.
  Interventions: Procedure: Corneal collagen crosslinking

INTERVENTIONS:
Procedure: Corneal collagen crosslinking — The patients will be submitted to corneal collagen crosslinking, that consists:
  Instillation of riboflavin eyedrop in the cornea for thirty minutes, and after, the patient will stay under the Crosslinking equipment, for more thirty minutes, also receiving riboflavin eyedrop.
  Other Names: Keratoconus.; Corneal collagen crosslinking.

SUMMARY:
The purpose of this study is to postpone the corneal transplantation in keratoconus and promote the stiffness of the cornea across the riboflavin-UVA corneal collagen crosslinking , and after, corneal ring surgery.

DETAILED DESCRIPTION:
Keratoconus is a progressive disease where cornea is thin and has a higher curvature.In early conditions, it may be corrected by glasses or contact lens.When these possibilities are not more possibles, it may be corrected by corneal ring surgery ore corneal transplantation depending your degree.

In this study, the patients with a degree of keratoconus on I or II, will be submitted to corneal collagen crosslinking and then a corneal ring surgery.

The corneal collagen crosslinking promote the stiffness of the cornea across the riboflavin-UVA irradiation, avoid the progression of the keratoconus.After three months of crosslinking, these patients will be submitted a corneal ring surgery.

These patients will be allowed by two years and various exams will realized them.

ELIGIBILITY:
Inclusion Criteria:

* Patients with keratoconus
* Patients that aren't using contact lenses
* Pachymetry more than 400Um
* Best visual acuity less or equal 20/30

Exclusion Criteria:

* Ocular surgeries before
* Other eye diseases
* Corneal curvature more than 65 dioptres

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Refractive data, visual acuity, topography patterns, pachymetry measurements. | Two years

SECONDARY OUTCOMES:
Anterior segment tomography data, corneal biomechanics, impression cytology. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Adimara C Renesto, MD, Principal Investigator — Federal University of São Paulo; Mauro S Campos, MD, Study Chair — Federal University of São Paulo; Marta F Sartori, MD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Mencucci R, Mazzotta C, Rossi F, Ponchietti C, Pini R, Baiocchi S, Caporossi A, Menchini U. Riboflavin and ultraviolet A collagen crosslinking: in vivo thermographic analysis of the corneal surface. J Cataract Refract Surg. 2007 Jun;33(6):1005-8. doi: 10.1016/j.jcrs.2007.03.021. PMID 17531694
- [Background] Coskunseven E, Kymionis GD, Tsiklis NS, Atun S, Arslan E, Jankov MR, Pallikaris IG. One-year results of intrastromal corneal ring segment implantation (KeraRing) using femtosecond laser in patients with keratoconus. Am J Ophthalmol. 2008 May;145(5):775-9. doi: 10.1016/j.ajo.2007.12.022. Epub 2008 Mar 4. PMID 18291344
- [Result] Wollensak G, Spoerl E. Collagen crosslinking of human and porcine sclera. J Cataract Refract Surg. 2004 Mar;30(3):689-95. doi: 10.1016/j.jcrs.2003.11.032. PMID 15050269
- [Derived] Renesto Ada C, Melo LA Jr, Sartori Mde F, Campos M. Sequential topical riboflavin with or without ultraviolet a radiation with delayed intracorneal ring segment insertion for keratoconus. Am J Ophthalmol. 2012 May;153(5):982-993.e3. doi: 10.1016/j.ajo.2011.10.014. Epub 2012 Jan 20. PMID 22265143